CLINICAL TRIAL: NCT02885363
Title: Prognosis of Isolated Left Ventricular Non-compaction in Adults
Acronym: NCVG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-20; 2011-A00987-34 (Other: ANSM)
Record Dates: First submitted 2016-08-17; First posted 2016-08-31 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Left Ventricular Non Compaction
MeSH Terms: interventions — Restraint, Physical; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with newly diagnosed Left Ventricular Non Compaction (Experimental): Patient newly diagnosed with Left Ventricular Non Compaction (diagnose < 6 months), confirmed by echocardiography associated or not with MRI, after centralized review
  Interventions: Other: Clinical examination; Other: Blood sample; Procedure: Echocardiography
- Patients with Idiopathic Dilated Cardiomyopathy (Active Comparator): Patient newly diagnosed with Idiopathic Dilated Cardiomyopathy (diagnose < 6 months), confirmed by echocardiography associated or not with MRI, after centralized review
  Interventions: Other: Clinical examination; Other: Blood sample; Procedure: Echocardiography

INTERVENTIONS:
Other: Clinical examination
Other: Blood sample
Procedure: Echocardiography

SUMMARY:
The main objective of this study is to clarify prospectively prognosis of patients newly diagnosed as carriers of a LVNC (incident cases) (i.e. without the occurrence of a survival of the following events: death, heart transplantation or hospitalization for cardiovascular complications). In a second time, prognosis factors will be identify in these patients with LVNC.

DETAILED DESCRIPTION:
Isolated Left Ventricular Non Compaction (LVNC) is a rare cause of cardiomyopathy supposed to result from the cessation of normal embryogenesis infarction, and characterized by persistent ventricular trabeculations prominent.

This is frequently a familial disease, but for which genetic characterization is still incomplete, and then requires the identification of new genes is desirable.

The prognosis of LVNC is uncertain, with a mortality rate reported in the literature ranging from 2 to 38%. Some series conclude that LVNC is a very severe heart disease, responsible for a high mortality, other that LVNC is frequently associated with a favorable prognosis. These series are however limited by the short duration of follow-up and the small number of patients included.

Between 2004 and 2006, a French registry LVNC, included 105 cases. It was found out that the LVNC was associated with a high rate of complications such as outbreaks of severe heart failure, need for heart transplantation, severe rhythm disorders, and embolic events. The prognosis of LVNC in France appears as pejorative:

1. - there is no evidence that prognosis is different from other forms of cardiomyopathies.
2. - the results of this register can be skewed by the inclusion of incident and prevalent cases (statistical survival bias).

Thus, a longer-term monitoring and the identification of relevant prognostic markers are imperative to better understand this rare disease and to improve the therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged over 18 years
* Presenting with Left Ventricular Non Compaction (LVNC, Group 1) or Idiopathic Dilated Cardiomyopathy (DCM, Group 2)
* At distance of an acute heart failure thrust (> 1 month)
* Newly diagnosed (less than 6 months)
* Diagnosis confirmed by echocardiography associated or not with a Magnetic Resonance Imaging (MRI) confirmed after central review
* Having signed informed consent form

Exclusion Criteria:

* Age <18 years
* Patients who were diagnosed more than 6 months ago (prevalent cases)
* Presence of an associated cardiac disease, including valvular, ischemic, or congenital disease
* Refusal to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2011-12-21 (Actual); Primary Completion 2015-10-23 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of death of cardiac origin | Up to 2 years
Occurrence of a cardiac transplantation | Up to 2 years
Occurrence of hospitalization due to cardiac event | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Hôpital de la Timone, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided